CLINICAL TRIAL: NCT03460379
Title: Bariatric Surgery and Pharmacokinetics Escitalopram: BAR-MEDS Escitalopram
Brief Title: Bariatric Surgery and Pharmacokinetics of Escitalopram
Status: Recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Volvat Medisinsk Senter Stokkan (Other); Namsos Hospital (Other); Alesund Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/1145k
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Obesity, Morbid
Keywords: Bariatric surgery; Gastrointestinal tract; Biological availability; Pharmacokinetics; Citalopram
MeSH Terms: conditions — Obesity, Morbid | interventions — Escitalopram; Citalopram

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Escitalopram — Patients are tested for their normal prescription escitalopram medication
  Other Names: Citalopram; Cytalopram

SUMMARY:
Changes to gastric pH, gastric emptying time, gastrointestinal transit-time or the pre-systemic metabolizing effect of enzymes secreted in the mucosa may all alter the pharmacokinetics of medicines. These factors are potentially influenced by bariatric surgery. Little is so far known about how gastric bypass and sleeve gastrectomy impacts the biological availability of medication. In this study the pharmacokinetic effects of bariatric surgery on escitalopram are investigated.

ELIGIBILITY:
Inclusion Criteria:

* Preparing to undergo gastric bypass or sleeve gastrectomy in Central Norway
* Being a Norwegian citizen

Exclusion Criteria:

* Having previously undergone resections in the GI-tract

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for bariatric surgery (gastric bypass or sleeve gastrectomy)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2016-11-02 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Escitalopram concentration in blood serum (area under curve (AUC)) | From baseline to 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Strømmen, MSc, Principal Investigator — St. Olavs University Hospital
Locations (1):
- St. Olavs University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schoretsanitis G, Strommen M, Krabseth HM, Helland A, Spigset O. Effects of Sleeve Gastrectomy and Roux-en-Y Gastric Bypass on Escitalopram Pharmacokinetics: A Cohort Study. Ther Drug Monit. 2023 Dec 1;45(6):805-812. doi: 10.1097/FTD.0000000000001114. Epub 2023 Jun 15. PMID 37363832